CLINICAL TRIAL: NCT03342144
Title: Observational Study of the Use of Venetoclax in Patients With Chronic Lymphocytic Leukemia (CLL) Under Real-Life Setting in Austria, Germany and Switzerland
Brief Title: Study of the Use of Venetoclax in Participants With Chronic Lymphocytic Leukemia (CLL) Under Real-Life Setting
Acronym: VeRVe
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P17-132
Record Dates: First submitted 2017-11-10; First posted 2017-11-14 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: Chronic Lymphocytic Leukemia (CLL); Cancer; Leukemia; venetoclax; rituximab; obinutuzumab; ABT-199; venclexta; venclyxto
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms; Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Participants Receiving Venetoclax: Participants with Chronic Lymphocytic Leukemia (CLL) receiving venetoclax.
- Participants Receiving Venetoclax + Rituximab: Participants with CLL receiving venetoclax in combination with rituximab.
- Participants Receiving Venetoclax + Obinutuzumab: Participants with CLL receiving venetoclax in combination with obinutuzumab.
- Participants Receiving Venetoclax + Ibrutinib: Participants with CLL receiving venetoclax in combination with ibrutinib.
- Participants Receiving Venetoclax + Acalabrutinib: Participants with CLL receiving venetoclax in combination with acalabrutinib.

SUMMARY:
An observational study to assess the effectiveness, health economic-relevant costs and participant reported outcomes in participants with Chronic lymphocytic leukemia (CLL) receiving venetoclax as a monotherapy or in combination with rituximab, obinutuzumab, ibrutinib, or acalabrutinib as prescribed at the discretion of the physician and in accordance with local clinical practice and label.

ELIGIBILITY:
Inclusion Criteria:

- Participant with chronic lymphocytic leukemia (CLL) who start venetoclax therapy can be included in the study if treated as specified in the local label for any specific line of treatment.

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with chronic lymphocytic leukemia (CLL) administering venetoclax per the local label.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-12-04 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Best Overall Response Rate (ORR) | Up to 12 months
  ORR is defined as the percentage of participants achieving partial response (PR) and complete response with incomplete regeneration of bone marrow (CRi) and complete response (CR) according to physician's assessment to therapy with venetoclax.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (70):
- Austria (4):
  - Universitaetsklinikum St. Poelten /ID# 221152, Sankt Pölten, Lower Austria
  - Medizinische Universitaet Graz /ID# 221155, Graz, Styria
  - Landeskrankenhaus Salzburg-Universitaetsklinikum der PMU (LKH) /ID# 221153, Salzburg
  - Hanusch Krankenhaus /ID# 221151, Vienna
- Germany (57):
  - Stauferklinikum Schwaebisch Gmuend /ID# 201518, Mutlangen, Baden-Wurttemberg
  - Onkologische Praxis /ID# 201545, Stuttgart, Baden-Wurttemberg
  - Schwarzwald-Baar-Klinikum /ID# 208176, Villingen-Schwenningen, Baden-Wurttemberg
  - MVZ am Klinikum Aschaffenburg Onkologie /ID# 201548, Aschaffenburg, Bavaria
  - Studienzentrum Aschaffenburg /ID# 204125, Aschaffenburg, Bavaria
  - Gemeinschaftspraxis Dr. Heinrich und Prof. Bangerter /ID# 200950, Augsburg, Bavaria
  - Drs. Tanzer, Chirca, Stoeberl /ID# 202613, Bad Reichenhall, Bavaria
  - Internistische Schwerpunktpraxen, Erlangen /ID# 200949, Erlangen, Bavaria
  - Onkologie Hof /ID# 201531, Hof, Bavaria
  - Praxis Dr. Stauch /ID# 202611, Kronach, Bavaria
  - VK&K Studien GbR /ID# 202614, Landshut, Bavaria
  - Haemato-Onkologie /ID# 205236, Munich, Bavaria
  - Praxis Dr. Kreher /ID# 202604, Bad Liebenwerda, Brandenburg
  - Praxis Dres. Kiehl/Stein /ID# 210052, Frankfurt (Oder), Brandenburg
  - MVZ f. Blut- u.Krebserkrankungen /ID# 206704, Potsdam, Brandenburg
  - Ambulantes Tumorzentrum Bremerhaven /ID# 224353, Bremerhaven, City state Bremen
  - Centrum fuer Haematologie und Onkologie Bethanien /ID# 206701, Frankfurt am Main, Hesse
  - MVZ Dres. Cordes & Partner /ID# 202598, Frankfurt am Main, Hesse
  - Klinikum Frankfurt Hoechst /ID# 210048, Frankfurt am Main, Hesse
  - Praxis Dres. Tebbe/Mayer /ID# 206730, Kassel, Hesse
  - Onkologische Kooperation Harz /ID# 201550, Goslar, Lower Saxony
  - OAZ Hannover /ID# 201538, Hanover, Lower Saxony
  - Onkolologische Praxis Oldenburg /ID# 202607, Oldenburg, Lower Saxony
  - MVZ der Paracelsus-Klinik /ID# 201541, Osnabrück, Lower Saxony
  - Med. Studiengesellschaft Nord West GmbH /ID# 201535, Westerstede, Lower Saxony
  - Praxis Dres. Plewe/Losem /ID# 202606, Neuss, North Rhine-Westphalia
  - Hämatologie und Onkologie /ID# 205247, Kaiserslautern, Rhineland-Palatinate
  - Praxis Dr. Klaproth/Cura /ID# 216413, Neunkirchen, Saarland
  - Onkozentrum Dresden /ID# 202599, Dresden, Saxony
  - BAG Freiberg-Richter, Jacobasch, Illmer, Wolf /ID# 201532, Dresden, Saxony
  - Luebecker Oncology Practice /ID# 200952, Lübeck, Schleswig-Holstein
  - Friedrich-Ebert-Krankenhaus GmbH /ID# 206206, Neumünster, Schleswig-Holstein
  - Praxis Dres. Krober/Stosiek /ID# 206729, Regensburg, State of Berlin
  - Caritas-Krankenhaus gGmbH /ID# 243212, Bad Mergentheim
  - MVZ Klinikum Mittelbaden GmbH /ID# 206207, Baden-Baden
  - Praxis für Hämatologie und Onkologie /ID# 241763, Berlin
  - Onkologische Schwerpunktpraxis /ID# 200953, Berlin
  - Praxis am Volkspark /ID# 243195, Berlin
  - Onkologie am Segelfliegerdamm /ID# 202603, Berlin
  - Pioh Dres. Draube & Partner /ID# 239507, Cologne
  - Praxis Dres. Prange-Krex/Mohm /ID# 210049, Dresden
  - St. Georg Klinikum Eisenach gemeinnützige GmbH (GKE) /ID# 250200, Eisenach
  - Praxis fuer interdisziplinaere Onkolologie und Haematologie /ID# 206999, Freiburg im Breisgau
  - MVZ Onkologie GmbH /ID# 212376, Hagen
  - onkomedic GbR /ID# 218354, Halle
  - OncoResearch Lerchenfeld GmbH /ID# 205237, Hamburg
  - Onkologische Gemeinschaftspraxis /ID# 205239, Hamburg
  - Evangelisches Krankenhaus Hamm /ID# 206703, Hamm
  - Studienzentrum am Raschplatz /ID# 250180, Hanover
  - Studienbüro Kamal und Dorn GBR /ID# 234105, Hanover
  - Klinikum Idar-Oberstein GmbH /ID# 210046, Idar-Oberstein
  - Praxis Fuchs/Koehler /ID# 243215, Langenhessen
  - Bruederkrankenhaus St. Josef Paderborn /ID# 202600, Paderborn
  - Onkologische Praxis GbR /ID# 206705, Porta Westfalica
  - Praxis Dres. Decker/Lakner/Leithäuser /ID# 206208, Rostock
  - Diakonieklinikum Schwaebisch Hall /ID# 206205, Schwäbisch Hall
  - MVZ am Schlossgarten GmbH /ID# 210043, Schwetzingen
- Switzerland (9):
  - Kantonsspital Aarau AG /ID# 210034, Aarau, Canton of Aargau
  - Spital Thun /ID# 233714, Thun, Canton of Bern
  - Luzerner Kantonsspital /ID# 210029, Lucerne, Canton of Lucerne
  - Réseau Hospitalier Neuchâtelois /ID# 227865, Neuchâtel, Canton of Neuchâtel
  - Kantonsspital St. Gallen /ID# 223037, Sankt Gallen, Canton of St. Gallen
  - KSW Kantonsspital Winterthur /ID# 211068, Winterthur, Canton of Zurich
  - EOC Ospedale Regionale di Bellinzona e Valli /ID# 208782, Bellinzona, Canton Ticino
  - Kantonsspital Münsterlingen /ID# 210035, Münsterlingen, Thurgau
  - Inselspital, Universitaetsspital Bern /ID# 210031, Bern

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schwaner I, Kuhn T, Losem C, Wolff T, Otremba B, Zaiss M, Hulsenbeck J, Famulla K, Nosslinger T, Rossi D. Low incidence of tumor lysis syndrome in elderly patients with chronic lymphocytic leukemia treated with venetoclax under real-world conditions: results from the prospective observational VeRVe study. Ann Hematol. 2024 Jun;103(6):2013-2020. doi: 10.1007/s00277-024-05638-7. Epub 2024 Feb 29. PMID 38421404
- See also: Related Info — http://www.rxabbvie.com/